CLINICAL TRIAL: NCT04916990
Title: Improving the Timeliness and Quality of Care for Rural Cancer Patients With Solid Tumors
Brief Title: Improving Care for Rural Patients With Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-2666.cc; P30CA046934 (NIH); R01CA254730-01 (NIH)
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer; Head and Neck Cancer; Thyroid Cancer; Cervical Cancer; Breast Cancer; Bladder Cancer; Colon Cancer; Rectum Cancer
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms; Thyroid Neoplasms; Uterine Cervical Neoplasms; Breast Neoplasms; Urinary Bladder Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARES Intervention (Active Comparator): All participants will complete surveys to assess Quality of Care and Patient Reported outcomes at baseline, 3 months and 6 months. The CARES intervention will include a maximum of 10 navigation and 10 counseling sessions delivered over approximately a 6- month period delivered by oncology nurse navigators and master's level counselors. Sessions will be scheduled to correspond with key transition points during treatment and may be held in person, virtually, or by phone.
  Interventions: Behavioral: CARES Intervention
- Usual Care (No Intervention): All participants will complete surveys to assess Quality of Care and Patient Reported Outcomes. Patients will receive a standardized list of resources.

INTERVENTIONS:
Behavioral: CARES Intervention — Nurse navigators and masters levels counselors will meet with participants up to 10 times each (10 navigation and 10 counseling) over a 6 month period. The number of sessions will be determined by the length of the patient's treatment. The timing of each session will be guided by a regular assessment to reduce the time from diagnosis to initiation of treatment and the time between subsequent treatments. Sessions will occur at key transition points during treatment to target the factors associated with treatment delays, reduced Quality of Care and poor Patient Reported Outcomes
  Arms: CARES Intervention

SUMMARY:
This study will assess if the CARES (Cancer Advocacy, Resources, Education and Support) intervention improves time to start of treatment after diagnosis and time to treatment completion for solid tumors (ex: lung, head, neck, thyroid, cervical, breast, bladder, colon, and rectal cancers) in rural patients.

DETAILED DESCRIPTION:
This is a randomized study. 320 participants will be enrolled to the CARES intervention or usual care arms. All participants will complete surveys to assess Quality of Care and Patient Reported outcomes at baseline, 3 months and 6 months. The CARES intervention will include a maximum of 10 navigation and 10 counseling sessions delivered over approximately a 6- month period delivered by oncology nurse navigators and master's level counselors. Sessions will be scheduled to correspond with key transition points during treatment and may be held in person, virtually, or by phone. Patients enrolled to the usual care arm will receive a standardized list of resources. Participation will last 6 months.

ELIGIBILITY:
Inclusion Criteria Assessed During Screening:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Male and female adults over 18 years old
4. English or Spanish speaking
5. Receives cancer treatment at UCH- Aurora, UCH-Highlands Ranch, UCHealth North, UCHealth South- UCHealth Memorial Hospital, UCHealth Parkview Hospital, San Juan Cancer Center, RMCC-Pueblo, SCL-St. Mary's, or Parkview Medical Center.
6. Resides in any of the rural counties served by the UCH-Aurora, UCH-Highlands Ranch, UCHealth North, UCHealth South- UCHealth Memorial Hospital, UCHealth Parkview Hospital, San Juan Cancer Center, RMCC-Pueblo, SCL-St. Mary's, VA, Huntsman Cancer Institute, or Parkview Medical Center with Rural-Urban Continuum Codes (RUCC) codes 4-9.
7. Diagnosed with lung cancer (LC): small cell lung cancer (SCLC), non-small cell lung cancer (NSCLC), using incident LC diagnosis according to the International Classification of Diseases for Oncology [ICD-O] codes: C34.0, C34.1, C34.2, C34.3, C34.8, C34.9, and C33.9, and other lung cancer variants
8. Stage of diagnosis for SCLC (limited vs. extensive), NSCLC (Stages 0, I, II, IIA, IIIB, IV), according to the American Joint Committee on Cancer Staging [AJCC] Tumor Node Metastasis [TNM] stages: I-IV)
9. Will receive the following types of breast, bladder, cervix, colon, rectum, lung, head-and-neck cancer treatments (surgery, radiation therapy, chemotherapy, or a combination of those modalities, including neoadjuvant and adjuvant therapy)
10. Diagnosed with head and neck cancer (HNC) using head and neck squamous cell carcinoma (HNSCC) ICD-O codes for the oral cavity (including lip; codes C00.0-C00.6, C00.8, C00.9, C02.0-C02.3, C02.8, C0.2.9, C03.0, C03.1, C03.9-C04.1, C04.8-C05.0, C06.0-C06.2, C06.8, and C06.9), the oropharynx (codes C01.9, C02.4, C05.1, C05.2, C5.8, C5.9, C09.0, C09.1, C09.8-C10.4, C10.8, C10.9, C14.0, C14.2, and C14.8), the hypopharynx (codes C12.9-C13.2, C13.8, and C13.9), and the larynx (codes C32.0- C32.3 and C32.8-C32.9) and histology codes for squamous cell carcinoma (SCC) or its variants (codes 8032, 8050, 8052, 8070-8075, and 8083-8084), and salivary gland cancer (code C07 and variants), and other head and neck cancer variants
11. Stage of diagnosis for HNC (Stages I, II, III, IV) according to the AJCC's TNM stages I-IV
12. Diagnosed with malignant neoplasm of thyroid gland, ICD-10 code: C73, and other thyroid cancer variants
13. Diagnosed with BC using malignant neoplasm of breast ICD-O codes for connective tissue of the breast, codes: C50.0, C50.1, C50.2, C50.3, C50.4, C50.5, C50.6, C50.8, C50.9, and other breast cancer variants.
14. Diagnosed with CC using malignant neoplasm of cervix uteri ICD-O codes: C53.0, C53.1, C53.8, C53.9 and other cervical cancer variants.
15. Diagnosed with CRC using colon and rectum malignant neoplasm ICD-O codes for colon (codes: C18, C18.1, C18.2, C18.3, C18.4, C18.5, C18.6, C18.7, C18.8, C18.9) and rectum (code C20), and other colon and rectum cancer variants.
16. Diagnosed with BLC using malignant neoplasm of ICD-O codes: C67.9 and other bladder cancer varients.

    Inclusion Criteria Confirmed via Baseline Survey:
17. Rural and medically underserved, defined as meeting the following criteria:

    * Rural: Resides in a rural county with a RUCC code 4-9 AND,
    * Underserved population who come from counties meeting any of the "health professional shortage areas" OR "Medically Underserved Areas/Populations" AND/OR
18. Uninsured: No health insurance (public or private insurance) AND/OR
19. Underinsured: (c.1) Public insurance (e.g., Medicaid, Medicare Part B exclusive, VA) (c.2) 10% or more of annual income is spent on out-of-pocket medical expenses

Exclusion Criteria Assessed During Screening:

1. Children under 18 years old
2. Individuals who do not speak English or Spanish
3. Individuals not receiving cancer treatment at UCH (Aurora, Highlands Ranch, UCHealth North, UCHealth Memorial Hospital), San Juan Cancer Center, RMCC-Pueblo, St. Mary's or Parkview Medical Center.
4. Diagnosed with primary cancer other than breast, bladder, cervix, colon, rectum, lung, and/or head-and-neck cancer or other type of cancer not listed in the inclusion criteria.
5. Diagnosed with a type of breast, bladder, cervix, colon, rectum, lung, and/or head-and-neck cancer listed under inclusion criteria but will not be treated at one of the collaborating hospital sites,
6. Has already initiated curative treatment for the current episode of cancer.

   Exclusion Criteria Assessed via Baseline Survey:
7. Individuals from vulnerable populations (e.g., inmates or on probation, homeless*, and pregnant*)
8. Decisionally-challenged with cognitive or personality impairment, suicidal ideation or intoxication (alcohol or drugs) at the time of consent or endorsed in baseline survey that interfere with ability to participate in the study.
9. Unable to hear (not including individuals who can hear with an auditory aid).*
10. Likely inability to track the individual over time (e.g. no permanent address at the time of consent) *Individuals who become homeless, pregnant, or lose their hearing or permanent address after they have consented and/or assigned to study condition may remain in the study until completion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to care | From study start to study end (6 months)
  Number of days from diagnosis to treatment initiation and number of days from treatment initiation to treatment completion

SECONDARY OUTCOMES:
Quality of Care | From study start to study end (6 months)
  Use Quality of Care (QOC) questionnaire to determine if CARES intervention results in favorable QOC experience
Patient Reported Outcomes | From study start to study end (6 months)
  Use Patient Reported Outcomes (PRO) questionnaire to determine if CARES intervention results in improvements in distress, adaptive coping, and tobacco use

CONTACTS AND LOCATIONS:
Overall Officials: Evelinn Borrayo, PhD, Principal Investigator — University of Colorado, Denver
Locations (14):
- United States (14):
  - University of Colorado Hospital, Aurora, Colorado
  - Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - SCL- St. Mary's Medical Center, Grand Junction, Colorado
  - VA Western Colorado Health Care System, Grand Junction, Colorado
  - Greeley Campus, Greeley, Colorado
  - Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - San Juan Cancer Center, Montrose, Colorado
  - Rocky Mountain Cancer Center, Pueblo, Colorado
  - UCHealth - Parkview medical Center, Pueblo, Colorado
  - Yampa Valley Medical Center, Steamboat Springs, Colorado
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No